CLINICAL TRIAL: NCT01142102
Title: A Multicentre Feasibility Study of Online Adaptive Image Guided Radiotherapy for Muscle Invasive Bladder Cancer
Brief Title: Feasibility of Online Adaptive Radiotherapy for Muscle Invasive Bladder Cancer
Acronym: BOLART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROG 10.01; ACTRN12610000711011 (Registry Identifier: Austalian New Zealand Clinical Trial Regisrty)
Record Dates: First submitted 2010-05-27; First posted 2010-06-11 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Bladder Cancer
Keywords: Bladder; Radiotherapy; Online; Adaptive
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Radiation Therapy
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — A radical dose of radiotherapy to be delivered to the entire bladder volume: 64Gy in 32 fractions over 6 weeks and 2 treatment days.
  * Conventional plan is used to deliver treatment for fractions 1 to 7 using a standard planning approach and a CTV to PTV margin of 1.5cm.
  * Adaptive plan is used to deliver treatment for fractions 8 through 32 using the same standard techniques as for fractions 1 to 7 but using one of three specific CTV volumes,namely: small, average or large. In all these cases the CTV to PTV margin is 0.7cm. Image guidance using a treatment unit based verification CT unit (Cone Beam CT or CT on Rails)based on soft tissue delineation is used to position the treatment fields and select the plan to best cover the CTV.

SUMMARY:
The principal objective of the trial is to test the hypothesis that Online Adaptive Radiotherapy for Muscle Invasive Bladder Cancer is feasible across multiple Radiation Oncology departments.

DETAILED DESCRIPTION:
This is a single-arm multicentre feasibility trial in which the primary aim is to determine the compliance rate of patients to online adaptive radiotherapy for muscle invasive bladder cancer over multiple Australian and New Zealand centres. The compliance rate is defined as the proportion of patients successfully completing treatment without a major protocol deviation.

Subject to the accrual being at least 40 patients in the first 2 years, accrual will continue until a total of 50 patients have been accrued. If this accrual target is not met, then consideration will be given to stopping the trial early due to poor accrual. Each patient will be followed-up until 2 years after the last patient's date of accrual. Assessments for toxicity and recurrence or progression will take place at four weeks after completion of treatment, then three monthly from the end of treatment for the first 12 months and then 6 monthly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Has provided written Informed Consent for participation in this trial
* Histologically confirmed muscle invasive bladder cancer.
* Transitional cell, squamous cell, adenocarcinoma or mixed histology. Stage T2-4 N0 M0.
* An ECOG performance status score of 2 or less (see appendices).
* Life expectancy greater than 6 months.
* Considered suitable for radical radiotherapy.
* Participants capable of childbearing are using adequate contraception.
* Radiotherapy must be able to be commenced within 12 weeks of surgery.
* Available for follow up.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Previous pelvic radiotherapy
* Previous cystectomy
* A small contracted bladder
* Unilateral or bilateral hip replacement
* Small cell histology
* Clinical or radiological evidence of nodal or distant metastases
* Presence of indwelling urinary catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Compliance with Online Adaptive Radiation Therapy process | From the start date of radiotherapy to the last day of radiotherapy treatment (approxiamately 6 weeks and 2 days)
  A patient is considered to be compliant if that patient completes treatment without experiencing a major protocol deviation

SECONDARY OUTCOMES:
Pattern of failure and competing risks analysis | From date of enrolment, every three months after RT untill 24 months, then 6 monthly until the end of the trial
  Patients will be assessed at baseline, weekly durning radiotherapy, 1 month post radiotherapy, then every three months until two years post radiotherapy.
Disease Free survival | From date of enrolment, every three months after RT untill 24 months, then 6 monthly until the end of the trial
  Patients will be assessed at baseline, weekly durning radiotherapy, 1 month post radiotherapy, then every three months until two years post radiotherapy.
Acute Toxicity of >/= grade 3 (NCI CTCAE version 4.0) of gastointestinal, diarrhoea, nausea, vomiting, colitis, proctitis, renal/genitourinary, cyctitis non-infective, haematuria, uinary frequency, urinary urgency and urinary retension. | From start date of radiotherapy and within 3 months of completion of radiation treatment
  Patients will be assesed at baseline, weekly durning radiotherapy, then at one month and three months post radiotherapy.
Quality of Life | Within 2 weeks prior to commencement of treatment, during the last week of treatment, 1 and 18 months after the completion of treatment.
  Patients will be assessed at baseline, on the last day of radiotherapy, at one month post radiotherapy, then at 18 months follow up.
Late normal tissue effects | Between 3 months and 3 years after the completion of radiation treatment
  Patients will be assessed at 3 monts post radiotherapy, then every 3 months until 2 years post radiotherapy.
Time to Local Bladder Failure | From date of enrolment to date of local bladder failure
  Patients will be assessed at baseline, weekly durning radiotherapy, 1 month post radiotherapy, then every three months until two years post radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Farshad Foroudi, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (12):
- Australia (10):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Mater Hospital, Brisbane, Queensland
  - Townsville Hospital, Douglas, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Peter MacCallum Cancer Centre - Box Hill, Melbourne, Victoria
  - Peter MacCallum Cancer Centre - Morrabbin, Melbourne, Victoria
  - Alfred Hospital, Prahran, Victoria
- New Zealand (2):
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Waikato

REFERENCES:
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au